CLINICAL TRIAL: NCT00338728
Title: Phase II Study of Letrozole (Femara) Plus Imatinib Mesylate (Gleevec) for Postmenopausal Patients With ER and/or PR Positive Metastatic Breast Cancer
Brief Title: Letrozole and Imatinib Mesylate in Treating Postmenopausal Participants With Estrogen or Progesterone Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0384; NCI-2018-01843 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2003-0384 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Estrogen Receptor Positive; KIT Positive; PDGFR Positive; Postmenopausal; Progesterone Receptor Positive; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: interventions — Imatinib Mesylate; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (imatinib mesylate, letrozole) (Experimental): Participants receive imatinib mesylate PO BID and letrozole PO QD for 8 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Imatinib Mesylate; Drug: Letrozole

INTERVENTIONS:
Drug: Imatinib Mesylate — Given PO
  Other Names: CGP 57148; CGP57148B; Gleevec; Glivec; STI 571; STI-571; STI571
Drug: Letrozole — Given PO
  Other Names: CGS 20267; Femara

SUMMARY:
This phase II trial studies the side effects and how well letrozole and imatinib mesylate work in treating postmenopausal participants with estrogen or progesterone positive breast cancer that has spread to other places in the body. Letrozole is an antihormonal drug used in the standard treatment of hormonal sensitive breast cancer. Imatinib mesylate is a drug that binds to certain proteins on the tumor cells and prevents them from further growth. Imatinib mesylate is thought to prevent the potential resistance to letrozole, which may make the letrozole more effective. Giving letrozole and imatinib mesylate may work better in treating participants with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of letrozole plus imatinib mesylate in patients with estrogen receptor (ER) and or progesterone receptor (PgR) positive metastatic breast cancer.

II. To determine the safety and tolerability of letrozole plus imatinib mesylate in patients with metastatic breast cancer.

III. To determine the time to disease progression and overall survival in patients with metastatic breast cancer who are treated with letrozole plus imatinib mesylate.

OUTLINE:

Participants receive imatinib mesylate orally (PO) twice daily (BID) and letrozole PO once daily (QD) for 8 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at 1 and 4 weeks and at 2, 4, 6, 9, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women able to comply with the protocol requirements with metastatic breast cancer, whose tumors are estrogen (ER) and/or progesterone (PgR) positive, defined by core biopsy immunohistochemistry with greater than 10% positive malignant epithelial cells
* Patients must have documented expression of either PDGFR or CD117 (c-kit) by immunohistochemistry
* Patients may have received tamoxifen in the adjuvant/neoadjuvant or setting. Patients may have previously received chemotherapy in the adjuvant/ neoadjuvant setting, though this is not required. Prior chemotherapy for metastatic breast cancer is allowed. Concomitant bisphosphonates are allowed for patients with bone metastases and who have another site of measurable disease
* Post menopausal status defined by one of the following: no spontaneous menses for at least 1 year, in women greater than or equal to 55 years spontaneous menses within the past 1 year in women greater than or equal to 55 years with postmenopausal gonadotrophin levels (luteinizing hormone [LH] and follicle stimulating hormone [FSH] levels greater than 40 IU/L ) or postmenopausal estradiol levels (less than 5 mg/dl) or according to the definition of "postmenopausal range" for the laboratory involved bilateral oophorectomy
* Performance status, Eastern Cooperative Oncology Group (ECOG) greater than or equal to 2
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as greater than or equal to 10 mm with conventional techniques. Bone disease only will not be accepted as measurable disease. Pleural or peritoneal effusions will not be accepted as measurable disease
* Absolute neutrophil count (ANC) = 1.5 x 10 to the 9th power/L
* Platelets greater than or equal to 100.0 x 10 to the 9th power/L
* Hemoglobin greater than 10.0 g/dL
* Creatinine less than 1.5 mg/dl
* Total (T.) bilirubin less than 1.5 x normal
* Aspartate aminotransferase (AST) less than 2.5 x normal
* A life expectancy of at least 6 months
* Localized radiotherapy, which does not influence the signal of evaluable lesion, is allowed prior to the initiation of imatinib mesylate. Patients must have recovered from the myelosuppressive effects of previous radiotherapy (at least 2-4 weeks)
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Prior treatment with Femara or Gleevec
* Uncontrolled endocrine disorders such as diabetes mellitus, confirmed hypo- or hyperthyroidism, Cushing's syndrome, Addison's disease (treated or untreated)
* Patients with unstable angina, or uncontrolled cardiac disease (e.g. class III or IV New York Heart Association's functional classification)
* Other concurrent malignant disease with the exception of cone-biopsied in situ carcinoma of the cervix uteri, or adequately treated basal or squamous cell carcinoma of the skin, or other curable cancers e.g. Hodgkin's disease or non-Hodgkin lymphoma (NHL), provided 5 years have elapsed from completion of therapy, and there has been no recurrence
* Concomitant treatment with steroids, e.g. glucocorticoids for indications other than cancer, except aerosol for obstructive airways diseases and steroid injection to the joints for treatment of inflammation
* Other investigational drugs within the past 3 weeks and the concomitant use of investigational drugs
* History of non-compliance to medical regimens and patients who are considered potentially unreliable
* Patients with known brain metastasis
* Patients with known chronic liver disease (i.e., chronic active hepatitis, and cirrhosis)
* Patients with known diagnosis of human immunodeficiency virus (HIV) infection
* Patients who received chemotherapy within 4 weeks (6 weeks for nitrosourea or mitomycin-C) prior to study entry, unless the disease is rapidly progressing
* Patients who previously received radiotherapy to greater than or equal to 25% of the bone marrow
* Patients who had a major surgery within 2 weeks prior to study entry

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2003-10-03 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Banu Arun, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from November 2003 to October 2008. The participating subjects must sign the consent document pertaining to the study and meet all the eligibility criteria as mentioned in the protocol, before initiating on the study treatment.
Pre-assignment Details: The study start date is the activation date which is October 2, 2003, but the first patient consented was on November 3, 2003.
Groups:
- Letrozole and Imatinib Mesylate: Imatinib mesylate 400 mg by mouth twice a day daily for 28 days and Letrozole 2.5 mg once a day daily for 28 days cycle.
Period: Overall Study
Arm/Group | Letrozole and Imatinib Mesylate
Started | 59
Completed | 45
Not Completed | 14
Not completed — Screen Failure | 14

BASELINE CHARACTERISTICS:
Arm/Group | Letrozole and Imatinib Mesylate
Number analyzed (Participants) | 45
Age, Continuous [Median (Full Range); unit: years] | 62.4 [41.4 to 82.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Among participants with CR or PR as the best overall response, duration of response (DOR) was defined as the time from which measurement criteria were met for CR or PR until the date of progression. Progression-free survival (PFS) was defined as the time from study enrollment to disease progression or death from any cause, whichever occurred first. PFS data were censored at the time of removal from study. Overall survival (OS) was defined as the time from study registration to death from any cause. Information on vital status was collected following study completion through July 23, 2018 and was used in the determination of OS. Among patients with SD as the best overall response, duration of SD was defined as the time from study enrollment to disease progression or removal from study.
Time Frame: From the registration until disease progression, death, unacceptable toxicity, or withdraw of study consent, whichever occurred first assessed up to 182 months
Population: Five participants was non evaluable due participants did not complete the first 2 cycles. (8 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Letrozole and Imatinib Mesylate
Number analyzed (Participants) | 45
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 5
  SD (including non-CR/Non-PD)>/=24 weeks | 16
  SD (including non-CR/Non-PD)</=24 weeks | 8
  Progressive Disease | 11
  Non-Evaluable | 5

2. Primary Outcome: Overall Survival of Participants
Description: This sample size would provide an estimate of the objective response rate (ORR) 95% confidence intervals for the ORR and CBR were calculated using the exact binomial method. Among patients with CR or PR as the best overall response, duration of response (DOR) was defined as the time from which measurement criteria were met for CR or PR until the date of progression. Progression-free survival (PFS) was defined as the time from study enrollment to disease progression or death from any cause, whichever occurred first. PFS data were censored at the time of removal from study. Overall survival (OS) was defined as the time from study registration to death from any cause. Information on vital status was collected following study completion through July 23, 2018 and was used in the determination of OS. Among patients with SD as the best overall response, duration of SD was defined as the time from study enrollment to disease progression or removal from study.
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Letrozole and Imatinib Mesylate
Number analyzed (Participants) | 45
months
  Progression-free survival (PFS) | 8.7 [3.8 to 11.4]
  Overall Survival (OS) | 44.3 [34 to 55.3]

ADVERSE EVENTS:
Time Frame: From the registration until disease progression, death, unacceptable toxicity, or withdraw of study consent, whichever occurred first assessed up to 182 months
Arm/Group | Letrozole and Imatinib Mesylate
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 14/45
Other Adverse Events (participants affected / at risk) | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Letrozole and Imatinib Mesylate (N=45)
Diarrhea (Gastrointestinal disorders) | 7
Fatigue (General disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Elevated bilirubin (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Letrozole and Imatinib Mesylate (N=45)
Nausea (Gastrointestinal disorders) | 19
Vomitting (Gastrointestinal disorders) | 17
Heartburn (Gastrointestinal disorders) | 6
Diarrhea (grade 2) (Gastrointestinal disorders) | 10
Constipation (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 2
Rectal bleeding (Gastrointestinal disorders) | 1
Edema (Investigations) | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 10
Headache (grade 2) (Nervous system disorders) | 1
Pain (Nervous system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 6
Leukopenia (grade2) (Blood and lymphatic system disorders) | 4
Anemia (Blood and lymphatic system disorders) | 11
Infection (Investigations) | 3
Fatigue (General disorders) | 23
ALT elevation (Investigations) | 2
AST elevation (Investigations) | 3
ALP elevation (Investigations) | 2
Stomatitis (grade 2) (Investigations) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3
Rash (grade 2) (Skin and subcutaneous tissue disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hypopigmentation (grade 2) (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Sensory neuropathy (grade 2) (Nervous system disorders) | 2
Alopecia (grade 2) (Investigations) | 1
Hot flashes (grade 2) (Reproductive system and breast disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2009-08-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT00338728/Prot_SAP_000.pdf